CLINICAL TRIAL: NCT04677972
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study to Evaluate the Safety and Efficacy of SPI-1005 in Meniere's Disease and Open Label Extension Study to Evaluate the Chronic Safety of SPI-1005
Brief Title: SPI-1005 for the Treatment of Meniere's Disease
Acronym: STOPMD-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sound Pharmaceuticals, Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPI-1005-351
Record Dates: First submitted 2020-06-08; First posted 2020-12-21 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2023-11

CONDITIONS: Meniere Disease; Ménière
Keywords: ebselen; hearing loss; tinnitus; vertigo; dizziness; SPI-1005
MeSH Terms: conditions — Meniere Disease; Hearing Loss; Tinnitus; Vertigo; Dizziness | interventions — ebselen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SPI-1005 400 mg BID (Experimental): Oral administration of SPI-1005 400 mg BID for 28 days, with 84-day followup
  Interventions: Drug: Ebselen
- Placebo (Placebo Comparator): Oral administration of matching placebo BID for 28 days, with 84-day followup
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ebselen — Glutathione peroxidase mimetic
  Other Names: SPI-1005
  Arms: SPI-1005 400 mg BID
Drug: Placebo — Matching placebo containing excipients
  Arms: Placebo

SUMMARY:
The study is a randomized, double-blind, placebo-controlled, multi-center clinical trial (RCT) with open-label extension study (OLE), of SPI-1005 in adult subjects with definite Meniere's disease with active symptoms within three months preceding study enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Adult males/females, 18-75 years of age at the time of enrollment.
* Diagnosis of definite Meniere's Disease by AAO-HNS Amended 2015 Criteria.
* Hearing loss of ≥30 dB at 250, 500, or 1000 Hz at study enrollment.
* At least two of three active symptoms (tinnitus; aural fullness; vertigo or dizziness) of Meniere's disease by AAO-HNS Amended 2015 Criteria, within 3 months of study enrollment.

Exclusion Criteria:

* Current, or within 60 days prior to study enrollment, use of IV ototoxic medications
* History of otosclerosis or vestibular schwannoma.
* History of significant middle ear or inner ear surgery in the affected ear.
* Conductive hearing loss with air-bone gap ≥15 dB, otitis media, or mixed hearing loss.
* Significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, neurological, or psychiatric disease.
* Current use or within 30 days prior to study enrollment systemic steroids.
* Current use or within 7 days prior to study enrollment intratympanic steroids.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2023-09-19 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 84 days
  Safety and tolerability assessed based on comparison of adverse events vs. placebo
Change in low frequency hearing thresholds measured by pure tone audiometry | 56 days
  Co-primary efficacy endpoint; assessment of hearing by pure tone audiometry
Change in Words-in-Noise Test score | 56 days
  Co-primary efficacy endpoint; assessment of word recognition by Words-in-Noise Test

SECONDARY OUTCOMES:
Change in tinnitus severity | 56 days
  Tinnitus Functional Index (0-100) where higher score is worse outcome
Change in tinnitus loudness | 56 days
  Tinnitus Functional Index Question #2 -- How Strong or Loud was your Tinnitus? (0-10) where higher score is worse outcome
Change in vertigo severity | 56 days
  Vertigo Symptom Scale (0-60) where higher score is worse outcome
Change in aural fullness | 56 days
  Aural Fullness Scale (0-10) where higher score is worse outcome
Change in dizziness | 56 days
  Dizziness Handicap Inventory (0-100) where higher score is worse outcome

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of Southern California, Los Angeles, California
  - House Clinic, Los Angeles, California
  - Sacramento Ear, Nose, & Throat, Roseville, California
  - George Washington University, Washington D.C., District of Columbia
  - ENT and Allergy Associates of Florida, Boca Raton, Florida
  - Indiana University, Indianapolis, Indiana
  - Kansas University Medical Center, Kansas City, Kansas
  - Advanced ENT & Allergy, Louisville, Kentucky
  - Piedmont Ear, Nose & Throat Associates, Winston-Salem, North Carolina
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kil J, Harruff EE, Longenecker RJ. Development of ebselen for the treatment of sensorineural hearing loss and tinnitus. Hear Res. 2022 Jan;413:108209. doi: 10.1016/j.heares.2021.108209. Epub 2021 Feb 19. PMID 33678494
- [Background] Kil J, Pierce C, Tran H, Gu R, Lynch ED. Ebselen treatment reduces noise induced hearing loss via the mimicry and induction of glutathione peroxidase. Hear Res. 2007 Apr;226(1-2):44-51. doi: 10.1016/j.heares.2006.08.006. Epub 2006 Oct 6. PMID 17030476
- [Background] Kil J, Lobarinas E, Spankovich C, Griffiths SK, Antonelli PJ, Lynch ED, Le Prell CG. Safety and efficacy of ebselen for the prevention of noise-induced hearing loss: a randomised, double-blind, placebo-controlled, phase 2 trial. Lancet. 2017 Sep 2;390(10098):969-979. doi: 10.1016/S0140-6736(17)31791-9. Epub 2017 Jul 14. PMID 28716314